CLINICAL TRIAL: NCT06100380
Title: Elaboration of a Prioritization Score for Pharmaceutical Interviews in Patients Treated With Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20162*
Record Dates: First submitted 2020-11-24; First posted 2023-10-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Thromboembolic Event
MeSH Terms: conditions — Thromboembolism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with Thromboembolic event and Hemorrhage group: patients who present a hemorrhage or a thromboembolic event
  Interventions: Other: Survey
- patients without Thromboembolic event and Hemorrhage: patients who don't present a hemorrhage or a thromboembolic event
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Questionnaire

SUMMARY:
Oral anticoagulants have a prominent place in the strategy of prevention and treatment of thromboembolic diseases, especially in patients with atrial fibrillation. However, a study conducted by the National Fund for Health Insurance (Caisse primaire d'Assurance maladie, CPAM) in 2017 among nearly 35,000 patients with non-valvular atrial fibrillation showed that one in five patients stopped their oral anticoagulant without medical advice for at least 60 days during the first year of treatment.

In our establishment, patients hospitalized in the Cardiology departments and treated with oral anticoagulants benefit from pharmaceutical interviews on their treatment before they return at home. This activity, which exists since November 2014, is based on a team consisting on a pharmacy student, supervised by a pharmacist trained in therapeutic education.

In order to secure the management of patients treated by oral anticoagulants and to answer the requirements of Certification, the investigators wish to extend the pharmaceutical interviews to all of hospital's healthcare services. However, the large number of patients concerned, the shorter hospital stays and the difficulties to organize collective sessions in front of the diversity of treatments and diseases are parameters to be taken into account in the development of this activity. The provision of a targeting tool for patients with high risk of thromboembolism and / or hemorrhage is a prerequisite for organizing this institutional approach to support patients on anticoagulants.

In this context, the investigators want to establish a prioritization score to identify patients on oral anticoagulants with a higher drug risk.

DETAILED DESCRIPTION:
Oral anticoagulants are represented by two classes: vitamin K antagonists (VKA) and non-VKA oral anticoagulants (DOAC). They have a prominent place in the strategy of prevention and treatment of thromboembolic diseases, especially in patients with atrial fibrillation. Their prescription continues to increase in France.

However, a study conducted by the National Fund for Health Insurance (Caisse primaire d'Assurance maladie, CPAM) in 2017 among nearly 35,000 patients with non-valvular atrial fibrillation showed that one in five patients stopped their oral anticoagulant without medical advice for at least 60 days during the first year of treatment.

In our establishment, patients hospitalized in the Cardiology departments and treated with oral anticoagulants benefit from pharmaceutical interviews on their treatment before they return at home. This activity, which exists since November 2014, is based on a team consisting on a pharmacy student, supervised by a pharmacist trained in therapeutic education.

In order to secure the management of patients treated by oral anticoagulants and to answer the requirements of Certification, he investigators wish to extend the pharmaceutical interviews to all of hospital's healthcare services. However, the large number of patients concerned, the shorter hospital stays and the difficulties to organize collective sessions in front of the diversity of treatments and diseases are parameters to be taken into account in the development of this activity. The provision of a targeting tool for patients with high risk of thromboembolism and / or hemorrhage is a prerequisite for organizing this institutional approach to support patients on anticoagulants.

In this context, the investigators want to establish a prioritization score to identify patients on oral anticoagulants with a higher drug risk. Case-control study was performed at University hospital of Reims.

ELIGIBILITY:
Inclusion Criteria:

* For the case-subjects:
* Patient hospitalized at the Reims university hospital
* Patient treated with an oral anticoagulant (vitamin K antagonist: VKA or non-VKA oral anticoagulant: DOAC) since at least one month
* Patient with a serious hemorrhage or a thromboembolic event.
* For the control-subjects:
* Patient hospitalized at the Reims university hospital
* Patient treated with an oral anticoagulant (vitamin K antagonist: VKA or non-VKA oral anticoagulant: DOAC) since at least one month
* Without a serious hemorrhage or a thromboembolic event.

Exclusion Criteria:

* Patient physically or mentally not able to express non-opposition or opposition to the study;
* Patient protected by law;
* Patient physically or mentally not able to answer the surveys;
* Patient hospitalized in the month preceding the inclusion;
* Patient discharged from hospital before having answering the surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected during their hospitalization at University hospital of Reims if they are treated with an oral anticoagulant.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Number of thromboembolic event in patients treated with an oral anticoagulant | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided